CLINICAL TRIAL: NCT04941898
Title: Adynovate Special Drug Use Result Survey (Perioperative Administration)
Brief Title: A Study of TAK-660 in Surgical Procedures for People With Hemophilia A.
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-660-5002; jRCT2031210173 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-06-25; First posted 2021-06-28 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — BAX 855

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAK-660 15-50 international units per kilograms (IU/kg): Participants will receive TAK-660 15-50 IU/kg slow intravenous injection every 8- 24 hours until the bleeding is resolved or wound healing.
  Interventions: Biological: PEGylated Recombinant Factor VIII

INTERVENTIONS:
Biological: PEGylated Recombinant Factor VIII — Polyethylene glycol (PEG)-ylated full-length recombinant FVIII (rFVIII)
  Other Names: TAK-660; BAX855; ADYNOVATE

SUMMARY:
This study is about a factor VIII medicine called Adynovate (TAK-660) used during surgery for people with hemophilia A who have low blood levels of factor VIII.

The aims of this study are as follows:

* To check for side effects from TAK-660.
* To check how well TAK-660 controls bleeding when used routinely during surgery and other invasive procedures such as tooth extractions.

The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

During the study, participants will receive infusions of TAK-660 during their hospital stay for surgery according to their clinic's standard practice. The study doctors will check for bleeds and side effects from TAK-660 from surgery until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participants with blood coagulation factor VIII (FVIII) deficiency who received this drug during surgery or treatment after the start date of this survey.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with blood coagulation factor VIII (FVIII) deficiency who received this drug during surgery or treatment after the start date of this survey.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60dd6d7def0b71001e743dff

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 10 investigative sites in Japan, from 30 June 2021 to 15 March 2024 .
Pre-assignment Details: Participants with coagulation factor VIII (FVIII) deficiency who received Recombinant FVIII PEGylated (ADYNOVATE) for surgery/procedure were enrolled. Participants received ADYNOVATE Intravenous Infusion as part of a routine medical care.
Groups:
- Recombinant FVIII PEGylated Intravenous Infusion: Participants with coagulation factor VIII (FVIII) deficiency received Recombinant FVIII PEGylated (ADYNOVATE) Intravenous Infusion for surgery/procedure as part of a routine medical care.
Period: Overall Study
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Started | 16
Completed | 15
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (17.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 30 Days
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 2

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Up to 30 Days
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 1

3. Primary Outcome: Number of Participants With Adverse Drug Reaction
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 30 Days
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 0

4. Primary Outcome: Number of Participants With Serious Adverse Drug Reaction
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Up to 30 Days
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 0

5. Primary Outcome: Number of Participants With Adverse Reactions Categorized as Inhibitor Development, Shock, or Anaphylaxis
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. Number of participants with adverse reactions categorized as inhibitor development, shock, or anaphylaxis was reported.
Time Frame: Up to 30 Days
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
Participants | 0

6. Secondary Outcome: Intraoperative Hemostatic Efficacy of Recombinant FVIII PEGylated Intravenous Infusion
Description: The number of surgeries with each rating on hemostatic efficacy was counted and the percentage was reported. Intraoperative hemostatic efficacy was assessed by following four rating and criteria. Excellent: Intraoperative blood loss was less than or equal to that expected for the type of procedure performed in a non-hemophilic population (≤100%)), Good: Intraoperative blood loss was up to 50% more than expected for the type: of procedure performed in a non-hemophilic population (101-150%), Fair: Intraoperative blood loss was more than 50% of that expected for the type of procedure performed in a non-hemophilic population (>150%) None: Uncontrolled hemorrhage that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy with study drug or other replacement therapy.
Time Frame: Day 1 (date of surgery)
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation. The number analyzed was the number of participants with data available for analysis.
Measure: Number; unit: percentage in total surgeries
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 14
percentage in total surgeries
  Excellent | 93.3
  Good | 6.7
  Fair | 0
  Poor | 0

7. Secondary Outcome: Postoperative Hemostatic Efficacy of Recombinant FVIII PEGylated Intravenous Infusion 1 Day After Surgery
Description: The number of surgeries with each rating on hemostatic efficacy was counted and the percentage was reported. Postoperative hemostatic efficacy 1 day after surgery was assessed by following four rating and criteria. Excellent: Postoperative hemostasis achieved with study drug was as good or better than that expected for the type of surgical procedure performed in a nonhemophilic population, Good: Postoperative hemostasis achieved with study drug was probably as good as that expected for the type of surgical procedure performed in a nonhemophilic population, Fair: Postoperative hemostasis with study drug was clearly less than optimal for the type of procedure performed but was maintained without necessitating rescue therapy with study drug or other replacement therapy, None: Participant experienced uncontrolled bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy with study drug or other replacement therapy.
Time Frame: 1 Day post-surgery
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation.
Measure: Number; unit: percentage in total surgeries
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
percentage in total surgeries
  Excellent | 56.3
  Good | 37.5
  Fair | 6.3
  Poor | 0

8. Secondary Outcome: Postoperative Hemostatic Efficacy of Recombinant FVIII PEGylated Intravenous Infusion at Completion of Perioperative Management
Description: Postoperative hemostatic efficacy at completion of perioperative management was assessed by following four rating and criteria. Excellent: Postoperative hemostasis achieved after Day 1 with study drug was as good or better than that expected for the type of surgical procedure performed in a non-hemophilic population, Good: Postoperative hemostasis achieved after Day 1 with study drug was probably as good as that expected for the type of surgical procedure performed in a non-hemophilic population, Fair: Postoperative hemostasis with study drug after Day 1 was clearly less than optimal for the type of procedure performed but was maintained without necessitating rescue therapy with study drug or other replacement therapy, None: Participant experienced uncontrolled bleeding after Day 1 that was the result of inadequate therapeutic response despite proper dosing, necessitating rescue therapy with study drug or other replacement therapy.
Time Frame: At completion of perioperative management (approximately 30 days after surgery)
Population: as for outcome 6
Measure: Number; unit: percentage in total surgeries
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
Number analyzed (Participants) | 15
percentage in total surgeries
  Excellent | 50.0
  Good | 43.8
  Fair | 6.3
  Poor | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Recombinant FVIII PEGylated Intravenous Infusion
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant FVIII PEGylated Intravenous Infusion (N=15)
Melaena (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Recombinant FVIII PEGylated Intravenous Infusion (N=15)
Insomnia (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04941898/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT04941898/SAP_001.pdf